CLINICAL TRIAL: NCT01847014
Title: AC-055-402: An Extension of AC-055-401, a Multi-center, Open-label, Single-arm, Phase 3b Study of Macitentan in Patients With Pulmonary Arterial Hypertension to Psychometrically Validate the PAH-SYMPACT Instrument
Brief Title: Clinical Study of Macitentan in Patients With PAH to Psychometrically Validate PAH-SYMPACT Instrument
Acronym: SYMPHONYext
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Protocol-defined criterion of macitentan availability achieved.
Sponsor: Actelion (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AC-055-402
Record Dates: First submitted 2013-05-02; First posted 2013-05-06 (Estimated); Results first posted 2018-08-22 (Actual); Last update posted 2018-08-22 (Actual); Status verified 2018-06

CONDITIONS: Pulmonary Arterial Hypertension
Keywords: Pulmonary Arterial Hypertension (PAH); psychometric instrument; PAH-SYMPACT
MeSH Terms: conditions — Pulmonary Arterial Hypertension | interventions — macitentan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Macitentan (Experimental): Macitentan tablet, dose of 10 mg, once daily.
  Interventions: Drug: Macitentan

INTERVENTIONS:
Drug: Macitentan — Macitentan tablet, dose of 10 mg, once daily.
  Other Names: ACT-064992

SUMMARY:
SYMPHONY Extension is an extension of AC-055-401, a multi-center, open-label, single-arm, Phase 3b study of macitentan in patients with Pulmonary Arterial Hypertension to psychometrically validate the PAH-SYMPACT instrument. The objective is to assess the long-term safety of macitentan in subjects with PAH beyond the treatment in the AC-055-401 study.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent prior to any study-mandated procedure.
* Patients with PAH who completed study AC-055-401
* Women of childbearing potential must:
* Have a negative urine pregnancy test at Visit 1 and agree to perform monthly serum pregnancy tests.
* Agree to use two methods of contraception from Visit 1 until 1 month after study drug discontinuation.

Exclusion Criteria:

* Patients who prematurely discontinued study drug in study AC-055-401
* Females who are lactating or pregnant (positive Visit 1 pregnancy test) or plan to become pregnant during the study
* Known hypersensitivity to macitentan or its excipients or drugs of the same class

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2013-09-01 (Actual); Primary Completion 2015-10-01 (Actual); Study Completion 2017-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alain Romero, MD, Study Chair — Actelion Pharmaceuticals US, Inc; Gary Palmer, MD, MBA, Study Chair — Actelion Pharmaceuticals US, Inc.
Locations (2):
- United States (2):
  - Kentuckiana Pulmonary Associates, Louisville, Kentucky
  - The Carl & Edyth Lindner Center for Research & Education at The Christ Hospital, Cincinnati, Ohio

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All sites activated on the SYMPHONY AC-055-401 clinical trial were invited to participate in this open-label extension study. Due to meeting the study closure milestone, defined as the marketing of Opsumit on 18 OCT 2013, only two sites received activation. Recruitment occurred between Quarter 2 2013 and Quarter 3 2015.
Pre-assignment Details: Subjects who completed the sixteen week treatment of macitentan on the SYMPHONY AC-055-401 clinical trial were eligible to enter this open-label extension study.
Period: Baseline Extension Visit
Arm/Group | Macitentan
Started | 4
Completed | 4
Not Completed | 0
Period: Completion of Extension Study
Arm/Group | Macitentan
Started | 4
Completed | 0
Not Completed | 4

BASELINE CHARACTERISTICS:
Population: A total of four participants enrolled directly from the parent clinical trial, SYMPHONY AC-055-401 (NCT01841762). There was only one arm associated with the Extension study.
Arm/Group | Macitentan
Number analyzed (Participants) | 4
Age, Categorical [Count of Participants; unit: Participants] — Participant population is Extension Analysis Set, a total of four patients. Age of patients recorded.
  Participants
    <=18 years | 0
    Between 18 and 65 years | 3
    >=65 years | 1
Age, Continuous [Mean (Full Range); unit: Years] — Participant population is Extension Analysis Set, a total of four patients. Subject's age was captured in the SYMPHONY AC-055-401 Screening visit.
  Years | 60.8 [55.0 to 66.5]
Sex: Female, Male [Count of Participants; unit: Participants] — Participant population is Extension Analysis Set, a total of four patients. Subject's sex was captured in the SYMPHONY AC-055-401 Screening visit.
  Participants
    Female | 4
    Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Participant population is Extension Analysis Set, a total of four participants.
  Participants
    Hispanic or Latino | 0
    Not Hispanic or Latino | 4
    Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Patient population is the Extension Analysis Set (EAS), a total of 4 participants.
  Participants
    American Indian or Alaska Native | 0
    Asian | 0
    Native Hawaiian or Other Pacific Islander | 0
    Black or African American | 1
    White | 3
    More than one race | 0
    Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Incident Rate of Adverse Events (AEs).
Description: Safety events are reported and documented as defined in study protocol from baseline to end of treatment period including safety follow-up visit.
Time Frame: From Visit 1 to Post-treatment safety follow-up visit (30 days after discontinuation of the study drug).
Population: Four participants represent the Extension Analysis Set, who transitioned from completion of SYMPHONY AC-055-401 to this open-label extension clinical trial.
Measure: Count of Participants; unit: Participants
Arm/Group | Macitentan
Number analyzed (Participants) | 4
Participants
  Participants with severe intensity AEs | 1
  Participants with AEs | 3

ADVERSE EVENTS:
Arm/Group | Macitentan
All-Cause Mortality (participants affected / at risk) | 0/4
Serious Adverse Events (participants affected / at risk) | 1/4
Other Adverse Events (participants affected / at risk) | 3/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Macitentan (N=4)
Chronic Obstructive Pulmonary Disease Exacerbation (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary Arterial Hypertension Exacerbation (Cardiac disorders) | 1 (1)
Pulmonary Hypertension Exacerbation (Cardiac disorders) | 1 (1)
Right Heart Failure (Cardiac disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Macitentan (N=4)
Hyperlipidaemia (Metabolism and nutrition disorders) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1)
Type 2 Diabetes Mellitus (Metabolism and nutrition disorders) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1)
Right Heart Failure (Cardiac disorders) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Chest Pain (General disorders) | 1 (1)
Pain In Jaw (Musculoskeletal and connective tissue disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Renal Impairment (Renal and urinary disorders) | 1 (1)
Chronic Obstructive Pulmonary Disease Exacerbation (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary Arterial Hypertension Exacerbation (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary Hypertension Exacerbation (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1)
Flushing (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any study-related publication written independently by investigators must be submitted to Actelion for review at least 30 days prior to submission for publication or presentation. Upon review, Actelion provide comments, and may also request alterations and/or deletions for the sole purpose of protecting its confidential information an/or patient rights. Neither the institution nor the investigator should permit publication during such a review period.